CLINICAL TRIAL: NCT02254148
Title: The Effect of Multiple Doses of BI 187004 on the Single Dose Pharmacokinetics of Cytochrome P450 Substrates (Caffeine, Warfarin, Omeprazole, Metoprolol and Midazolam) and a P-glycoprotein Substrate (Digoxin) Administered Orally in an Open-label, One-sequence Trial in Healthy Subjects
Brief Title: The Effect of BI 187004 on the Pharmacokinetics of Cytochrome P450 Substrates (Caffeine, Warfarin, Omeprazole, Metoprolol and Midazolam) and a P Glycoprotein Substrate (Digoxin)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1307.19; 2013-005029-22 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam; Caffeine; Digoxin; Warfarin; Omeprazole; Metoprolol

ARMS (1):
- Treatment (Experimental): single dose of CYP 450 substrates and a P-gp substrate + multiple doses of BI 187004
  Interventions: Drug: midazolam; Drug: caffeine; Drug: digoxin; Drug: warfarin; Drug: omeprazole; Drug: BI 187004; Drug: metoprolol

INTERVENTIONS:
Drug: midazolam — single dose of midazolam given as oral solution (day 1 of visits 2 and 3)
Drug: caffeine — single dose of caffeine given as tablets (day 1 of visits 2 and 3)
Drug: digoxin — single dose of digoxin given as tablets (day 3 of visits 2 and 3)
Drug: warfarin — single dose of warfarin given as tablets (day 1 of visits 2 and 3)
Drug: omeprazole — single dose of omeprazole given as tablet (day 1 of visits 2 and 3)
Drug: BI 187004 — multiple doses of BI 187004 given as tablets (day 7-12 of visit 2 and day 1-6 of visit 3)
Drug: metoprolol — single dose of metoprolol given as tablets (day 1 of visits 2 and 3)

SUMMARY:
To assess the influence of BI 187004 on kinetics of cytochrome P450 (CYP) and P glycoprotein (P-gp) probe drugs as a means of predicting drug-drug interactions.

ELIGIBILITY:
Inclusion criteria:

1. healthy male subjects
2. age of 18 to 55 years
3. body mass index of 18.5 to 29.9 kg/m2
4. Subjects must be able to understand and comply with study requirements

Exclusion criteria:

1. Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease judged as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
AUC0-tz (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) for probe substrates | up to 143 hours postdose
Cmax (Maximum measured concentration of the analyte in plasma) for probe substrates | up to 143 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1307.19.1 Boehringer Ingelheim Investigational Site, Biberach, Germany